CLINICAL TRIAL: NCT05648370
Title: Liquid Biopsy in Advanced Oligometastatic NSCLC Receiving Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LB4S
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-07

CONDITIONS: Non-small Cell Lung Cancer; Oligometastatic Disease
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Every ctDNA test will take 20ml peripheral blood for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- oligometastatic disease: Dynamic blood samples before and after surgery and tissue samples from oligometastatic NSCLC undergone surgery will be obtained for exploratory analysis.
  Interventions: Genetic: ctDNA testing and whole exome sequencing

INTERVENTIONS:
Genetic: ctDNA testing and whole exome sequencing — Blood samples will be obtained for ctDNA testing and tumor tissue for whole exome sequencing.

SUMMARY:
A prospective, observational study that assesses the clinical feasibility of ctDNA-based liquid biopsy in patients with oligometastatic NSCLC receiving surgery.

DETAILED DESCRIPTION:
60 eligible patients will be enrolled. Dynamic blood samples before and after surgery and tissue samples will be obtained for exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained from patients and ability for patients to comply with the requirements of the study；
* Patients must be a man or woman of more than 18 years;
* ECOG PS ≦1；
* The function of the organs was evaluated by the surgeon to tolerate local surgical treatment；
* The classification was evaluated as simultaneous oligometastases at initial treatment or oligoresidual/oligoprogression/oligorecurrence after induction therapy; [Define: Initial treatment of simultaneous oligometastases: without systemic treatment, at the time of diagnosis, up to 5 metastases and up to 3 organs were involved, excluding pleural metastases or myeloid metastases.

Oligoresidual after induction therapy: after systemic therapy, distant metastases were stable or reduced, primary lesions were stable or reduced, PET/CT metabolism was reduced, and no more than 5 residual lesions and no more than 3 organs were involved.

Oligoprogression after induction therapy: After systemic therapy, some lesions were stable or reduced, while some original lesions were larger than before.

Oligorelapses after induction therapy: after systemic therapy, systemic lesions were stable or reduced, and new local lesions appeared.]

* Lesion evaluation can be surgically removed. [Definition of operable resection: the lesion is limited and can be completely removed through surgery as assessed by the surgeon, with no significant impact on postoperative quality of life. Pulmonary surgical procedures include lobectomy, segmental resection and wedge resection. Pneumonectomy is not included.]

Exclusion Criteria:

* Patients with a confirmed or suspected autoimmune disease;
* Patients with a history of human immunodeficiency virus (HIV) positive or acquired immunodeficiency syndrome (AIDS);
* Patients with a history of any arterial thrombosis within 6 months and history of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolism within 3 months;
* Patients with any unstable systemic disease (eg, active infection, high-risk hypertension, unstable angina, congestive heart failure, etc.);
* Patients with a history of other malignancies in the past 5 years;
* Patients identified by the investigators patients with contraindications to local treatment;
* Patients with serious mental illness;
* Patients who cannot sign informed consent;
* Patients who cannot be followed up as scheduled;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IV NSCLC patients with oligometastases at initial diagnosis or oligoresidual or oligoprogression or oligorelapses after systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Association between perioperative ctDNA-MRD characteristics and rogression-free survival | 2-year PFS
  To explore the potential association among perioperative ctDNA-MRD characteristics and rogression-free survival within 2 years.
Construction of a survival-prediction model | Through study completion, up to 5 years
  The survival-prediction model based on clinicopathological and genomic characteristics.

SECONDARY OUTCOMES:
Association among ctDNA status before surgery, systemic treatment times, and survival | Through study completion, up to 5 years
  To explore the potential association among plasma ctDNA status surgery, systemic treatment time duration, PFS and OS.
Genomic characteristics and clonal evolution after systemic treatment | Through study completion, up to 5 years
  Using whole-exome sequencing to identify genomic characteristics and clonal evolution after systemic treatment
Potential drug-resistance mechanism identified by plasma ctDNA | Through study completion, up to 5 years
  Using plasma ctDNA-MRD to identify the potential drug-resistance mechanism.
Assess whether ctDNA-MRD is associated with radiological and pathological response after systematic therapy before surgery | 60 patients underwent surgery
  Association among perioperative ctDNA-MRD characteristics, imaging response, and pathological response.
Heterogeneity in Genomic and transcriptome between primary and metastatic tumors | 60 patients underwent surgery
  Using whole-exome sequencing and whole transcriptome sequencing to identify genomic and transcriptome heterogeneity between primary and metastatic tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Zhao Zhong, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China